CLINICAL TRIAL: NCT03658837
Title: Functional Outcome Following Ivor-Lewis Oesophagectomy
Brief Title: Gastrointestinal Functional Outcome Ivor Lewis
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE ID 107692
Record Dates: First submitted 2018-07-13; First posted 2018-09-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ivor Lewis Oesophagectomy — Patients who underwent Ivor-Lewis Oesophagectomy for cancer of oesophagus

SUMMARY:
This study focuses on the prevalence of functional complications and their impact on QOL in patients who underwent an Ivor Lewis Oesophagectomy.

This study will assess the prevalence of gastrointestinal symptoms and QOL from beyond the first year following surgery up to 5 years. The aim is to determine whether gastrointestinal side effects and QOL are compromised in the long-term.

This study will also explore in details, the impact of surgery on their quality of life and gastro intestinal symptoms that patients has experienced post operatively.

DETAILED DESCRIPTION:
Oesophago-gastric (OG) cancer is the fifth most common malignancy in the United Kingdom, affecting approximately 16,000 people each year. Although surgery offers the best prospect for potential cure of OG cancers, radical treatment may result in increased treatment relate mortality, high treatment-induced morbidity, and reduced quality of life. Traditionally, many centres managing OG cancers focused on mortality and morbidity as their key outcome measures. However, a growing body of opinion considers that a measure of broader effects of ill health and treatment on the patients quality of life (QOL) is necessary. Such considerations are important as it is questionable if patients are subjected to treatment merely to offer them a few extra months of life, particularly if this is at the expense of quality of life. These includes physical, functional, social and physiological aspects of life.

More than half of the operated patients will develop significant functional disorder after surgery affecting QOL. The most common problems observed are dysphagia, dumping syndrome, delayed gastric emptying, and reflux. These functional disorder are not always detected immediately post operatively, but may become more troublesome as time goes by.

The purpose of this study is

* to evaluate mid to long term HRQL in patients that underwent Ivor Lewis esophagectomy (ILE) with gastric pull-up in Royal Leicester Infirmary with minimum of 12 months follow up and up to 5 years.
* to identify clinical factors influencing quality of life post operatively.
* explore patients' experiences of their quality of life and how they handle their new life situation from a long-term perspective after oesophagectomy The outcome of this study would benefit both surgeons and patients in terms of pre-operative counselling and planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Ivor Lewis Oesophagectomy in Leicester Royal Infirmary with minimum follow up of 12 months.
* Age more than 18

Exclusion Criteria:

* Disease recurrence within the follow up period
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent Ivor Lewis oesophagectomy with lymphadenectomy for oesophageal cancer will be selected from our database at the Department of Surgery, Leicester Royal Infirmary. These include patients from Leicestershire and Northamptonshire treated at the Leicester Royal Infirmary. Mid to long term survivors operated in our institution with a follow up of at least 12 months will be identified from our database to be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Quantitative Assessment using EORTC QLQ-C30 (version 3.0) | Beyond 12 months up to 5 years
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL,but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quantitative Assessment using EORTC QLQ-OES-24 | Beyond 12 months up to 5 years
  EORTC QLQ-OES-24 is a 24-item esophageal cancer-specific questionnaire supplementing EORTC QLQ-C30 with information about disease and treatment-related symptoms and side effects, dysphagia, nutrition, and social and emotional effects of esophageal cancer.
  Scale scores will be calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems

SECONDARY OUTCOMES:
Qualitative analysis | Beyond 12 months up to 5 years
  Interviews will be conducted with up to 15 participants and their carers and qualitative analysis of interviews will be performed

CONTACTS AND LOCATIONS:
Overall Officials: DAVID J BOWREY, MD, Study Director — University Hospitals, Leicester
Locations (1):
- Leicester Royal Infirmary, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03658837/Prot_000.pdf